CLINICAL TRIAL: NCT03463967
Title: Controlled Trial on the Effect of Tomato Products in Obese Children With Non Alcoholic Fatty Liver Disease
Brief Title: Effects of Tomato Products in Children With NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Iorio, Chief of the Pediatric Hepathology Unit, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TD1016
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: NAFLD
Keywords: nonalcoholic steatohepatitis; obesity; dyslipidemia; diet; children; adolescents
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Dyslipidemias | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycopene supplemented (Active Comparator): Energy-restricted diet supplemented with lycopene-enriched tomato juice
  Interventions: Dietary Supplement: Lycopene-enriched tomato juice; Other: Energy-restricted diet
- Calories Restricted (Sham Comparator): Energy-restricted diet
  Interventions: Dietary Supplement: Lycopene-enriched tomato juice; Other: Energy-restricted diet

INTERVENTIONS:
Dietary Supplement: Lycopene-enriched tomato juice — Energy-restricted diet supplemented with Lycopene-enriched tomato juice
  Other Names: TOMATO
Other: Energy-restricted diet
  Other Names: DIET

SUMMARY:
CONTROLLED TRIAL ON THE EFFECT OF TOMATO PRODUCTS IN OBESE CHILDREN WITH NON ALCOHOLIC FATTY LIVER DISEASE

Aim of the study To evaluate the effect of the addition of a daily dose of lycopene enriched tomato sauce on the progress of NAFDL in obese children.

Participants Children with obesity referred to the Hepatology unit of Dept.of Pediatric Clinic of the University Federico II of Naples. Diagnosis of NAFLD is made on the presence of fatty liver at ultrasound examination, with or without hypertransaminasemia.

Patients are eligible on the basis of:

* Age 4-14 years
* BMI > 85°percentile
* Liver Steatosis evaluated as mild, moderate or severe by US (hyperechogenic liver tissue compared with the adjacent kidney cortex)

Patients are excluded on the basis of:

* Liver disease
* Diabetes or manifest metabolic alterations
* Associated diseases Informed consent is obtained from the parents of the participating children. Sample size estimation To provide an 80% power to detect a 25% or greater relative shift of outcome variables, with a first degree error of .05 a sample of 50 cases is estimated in a cross over trial.

Study design This is a randomized, crossover, one side open trial with blinded outcome evaluation. A statistician who is not otherwise involved in the trial generated the randomized assignment sequence. At the enrollment all participants received a low carotenoids diet for two weeks (wash out), then children are assigned to the first intervention for 8 weeks, and subsequently, in the crossover phase, they are switched to the second intervention for the next 8 weeks. No wash out is planned between the two treatments.

Interventions

1. Supplemented diet: 100 gr/day of Lycopene enriched tomato products (weekly average)
2. Control diet: ordinary healthy diet, with no special encouragement to eat carotenes products All children are put on a 'mediterranean style' diet, with a controlled amount of calories: a dedicated dietitian for the whole study, irrespective of the treatment, checked their diet twice a week.

At beginning (T0) and at the end of each treatment (T1 and T2) all patients underwent anthropomorphic measurements, including weight, height, waist, abdomen and hips circumferences. BMI and its standard deviation score are calculated.

Regardless of group assignment, all participants are seen by a hepatologist at the end of each intervention and checked for liver steatosis, by US. Fasting blood samples are collected at beginning (T0) and at the end of each treatment (T1 and T2) to evaluate IR (assessed by HOMA), transaminases levels, lipids profile, oxidative state (assessed by antioxidant enzymes activity, serum levels of MDA and carbonylated proteins), inflammatory state (by cytokines serum levels, typing of lymphocytes subpopulations, metabolism of lymphocytes).

Data collection are performed in a partially blind fashion: the statistician performing data analysis is blind to treatment.

Outcomes: The primary outcome is reduction of the liver steatosis estimated by US Scan, according to the following parameters: parenchyma echogenicity (compared with that of the cortical of the right kidney), far gain attenuation, diaphragm blurring. steatosis.

Secondary outcomes is reduction in Insulin resistance, Oxidative state, Inflammatory state.

Statistical Analysis Data are inspected for normality and paired t-test (before/after) of each phase of the trial are performed when appropriate. The Median % change of each variable between the values at Time 8 and 16 weeks and values at enrollment are also looked. Ordinal logistic regression analysis, hierarchical, mixed model with adjustment variables are adopted to estimate the size of the effect.

The study is approved by the Ethical Committee of University Federico II of Naples.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-14 years
* BMI > 85°percentile
* Liver Steatosis evaluated as mild, moderate or severe by US (hyperechogenic liver tissue compared with the adjacent kidney cortex)

Exclusion Criteria:

* Liver diseases
* Diabetes or manifest metabolic alterations
* Associated diseases

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of liver steatosis | Baseline and 16 weeks
  The presence and severity of liver steatosis are graded by using the following criteria:
  2. The presence of hyperechogenic liver tissue (compared with the adjacent kidney cortex) with fine and tightly packed echo targets and of normal beam penetration with normal visualization of diaphragm and portal vein borders is considered as mild steatosis.
  3. The moderate and diffuse increase of echo intensity with decreased beam penetration (with slightly decreased visualization of diaphragm) associated with a decrease in visualization of silhouetting of the portal vein borders is considered as moderate steatosis.
  4. The marked increase in echoes intensity with no visualization of portal vein border, obscured diaphragm and posterior portion of the right lobe, and reduced visibility of kidney is considered as severe steatosis.
Reduction in BMI | Baseline and 16 weeks
  Standard methods of evaluation

SECONDARY OUTCOMES:
Reduction in ALT serum level | Baseline and 16 weeks
  Standard method of evaluation
Improvement of inflammatory state | Baseline and 16 weeks
  Evaluation of serum levels of standard markers of inflammation (CRP, ferritin); cytokines profiling, lymphocyte typing
Amelioration of oxidative state | Baseline and 16 weeks
  Evaluation of activity of serum antioxidant enzymes and markers of oxidative stress (MDA, Carbonylate proteins, oxidized LDL)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Iorio, Principal Investigator — University Federico II of Naples
Locations (1):
- Unit of Hepatology-Dept. of Pediatric Clinic, Naples, Italy

IPD SHARING:
Plan to Share IPD: No